Form M0345



Consent to Participate in a Research Study ADULT: 3<sup>rd</sup> Party Consent Form

Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

## AUDIO-RECORDING RELEASE FORM

We are conducting a research study where we will be audio-recording primary care clinical encounters between consenting DUHS clinicians and their enrolled patients. If you are in the room at the time of these recordings, it is possible that your voice will be on the audiotape.

- We will ask you if you are a member of the participating clinicians' staff, a student, or a visiting clinician.
- We will not be able to edit the recordings to remove your voice.
- These audio-recordings are uploaded to a password protected secure server or stored in a locked file cabinet in the offices of the Dr. Sarah Wilson and Dr. Laura Svetkey can only be accessed by authorized study staff.

We are asking you to sign this release form to acknowledge that you have been informed of the audio-recording taking place while you are in the room.

## STATEMENT OF CONSENT

"I have read and understand the foregoing and I consent to the use of my voice as specified for the above-described purpose. I further understand that no royalty, fee or other compensation of any character shall become payable to me by Duke University Health System or any of its affiliates for the use of my voice."

| Signature of Individual | Date |
|------------------------------|------|
| Divided Nove a Chadical dead | |
| Printed Name of Individual | |
| Signature of Study Staff | Date |